CLINICAL TRIAL: NCT01616212
Title: Early Intervention for Minors in Possession of Alcohol/Drugs: A Feasibility Study
Acronym: MAST1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA-12-033
Record Dates: First submitted 2012-05-29; First posted 2012-06-11 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Substance Use Disorder; Delinquency
Keywords: Teens; Parenting; Substance Abuse; Treatment Efficacy
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TX1 (Experimental): Motivational Enhancement Therapy for adolescents, Parenting Wisely for parents
  Interventions: Other: Motivational Enhancement Therapy /Adol and PW for parents
- TX 2 (Experimental): Motivational Enhancement Therapy for adolescents
  Interventions: Other: Motivational Enhancement Therapy for adolescents
- TX3 (Experimental): Drug Education for adolescents, Parenting Wisely for parents
  Interventions: Other: Drug Education for adolescents, Parenting Wisely for parents
- TX4 (Experimental): Drug Education for adolescents
  Interventions: Other: Drug Education for adolescents

INTERVENTIONS:
Other: Motivational Enhancement Therapy /Adol and PW for parents — Motivational Enhancement Therapy for adolescents, Parenting Wisely for parents
  Other Names: MET / PW
  Arms: TX1
Other: Motivational Enhancement Therapy for adolescents — Motivational Enhancement Therapy for adolescents
  Other Names: MET
  Arms: TX 2
Other: Drug Education for adolescents, Parenting Wisely for parents — Drug Education for adolescents, Parenting Wisely for parents
  Other Names: EDUC / PW
  Arms: TX3
Other: Drug Education for adolescents — Drug Education for adolescents
  Other Names: EDUC
  Arms: TX4

SUMMARY:
The purpose of this study is to evaluate two brief, sustainable interventions for a sample of 280 adolescents charged with an initial drug-related offense: Motivational Enhancement Therapy (MET) intervention for youth and the Parenting Wisely (PW) intervention for parents. Families are assessed for adolescent substance use, HIV-risk, recidivist substance-related offenses, treatment entry, and other areas of individual and family functioning.

It is expected that the combined MET+PW interventions will be more effective than a treatment-as-usual intervention (drug education group) for adolescents with parents not participating in PW.

DETAILED DESCRIPTION:
Illicit substance use and related problems among adolescents has been consistently high over the past decade and remains one of the most pressing public health concerns in the United States. The objective of this study is to conduct a pilot investigation of the feasibility and effectiveness of two brief empirically based treatments for adolescent substance abuse when implemented as early interventions for youth arrested and charged with first- or second-offense possession of alcohol or drugs. The two examined interventions are Motivational Enhancement therapy (MET) and Parenting Wisely (PW).

Over a one-year period, 280 adolescents and their parents will be referred to the study by the Juvenile Justice Centers in two Oregon counties within the Portland metro area. Families will be randomized to one of four intervention conditions; youth will receive either MET or a drug education intervention (EDUC), and the PW intervention for parents is present or absent. Participants will be assessed for adolescent substance use, HIV-risk, recidivist substance-related offenses, treatment entry, and other areas of individual and family functioning at intake and at 3- and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. 13 - 17 years of age
2. Referral for a 1st or 2nd Minor in Possession (Alcohol) or Less Than an Ounce (Marijuana) offense
3. Adolescents living at home with at least one parent willing to participate in the study
4. Adolescents with sufficient English-language ability to permit participation in the interventions
5. Parent(s) with sufficient English- or Spanish-language ability to complete the English- or Spanish-language versions of PW and the assessment

Exclusion Criteria:

1. Evidence of psychotic or organic state of sufficient severity to interfere with understanding study procedures
2. Danger to self and/or services other than outpatient treatment are required

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Adolescent Substance Use and Related Problems | Change from Baseline at 6 months
  The questionnaire used is called the Time Line Follow Back.

SECONDARY OUTCOMES:
Dysfunctional Discipline Practices | Change from Baseline at 6 months
  The questionnaire used to obtain this information is called Parenting Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Hops, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Portland, Oregon, United States